CLINICAL TRIAL: NCT03745521
Title: An International, Multicenter, Prospective, Longitudinal Observational Study for Patient With X-linked Hypophosphatemic Rickets/Osteomalacia
Brief Title: Study of Longitudinal Observation for Patient With X-linked Hypophosphatemic Rickets/Osteomalacia in Collaboration With Asian Partners
Acronym: SUNFLOWER
Status: Active, not recruiting | Type: Observational
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SUNFLOWER; UMIN000031605 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2018-11-06; First posted 2018-11-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: X-Linked Hypophosphatemia
Keywords: XLH
MeSH Terms: conditions — Familial Hypophosphatemic Rickets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- X-linked Hypophosphatemia (XLH): Hypophosphatemic Rickets/osteomalacia
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Through observation of patients with X-linked hypophosphatemic rickets/osteomalacia (XLH) for up to 10 years, the study intends to collect data that allow achievement of the following objectives:

1. To determine medical characteristics of the disease and the disease process
2. To determine physical and psychological burden on patients as well as economic burden
3. To assess the efficacy and safety of the treatment of the disease

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet at least one of the following:

  1. Documented PHEX gene mutation
  2. Documented PHEX gene mutation in at least one family member with X-linked genetic relationship
  3. Documented FGF23 >30 pg/mL
* Typical clinical findings of rickets/osteomalacia
* Written informed consent obtained from patients aged >=18 years or from parents or legally acceptable representatives of patients aged <18 years

Exclusion Criteria:

* Participation in any clinical study (trial) at the time of informed consent
* Any patient whose participation in the study is considered inappropriate by the investigator or the subinvestigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with XLH independent of treatment regimen
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Height | After enrollment, patients will be observed annually or every 2 years for up to 10 years.
  Height in centimeters
The 6-Minutes Walking Test | After enrollment, patients will be observed annually for up to 10 years.
  The 6-Minutes Walking Test performed according to International Guidelines, will be measured as distance in meters.
Timed Up and Go Test(TUGT) | After enrollment, patients will be observed every 2 years for up to 10 years.
  The time required for each patient to do the TUGT will be recorded: Stand up from sitting in a chair, walk 3 meters, turn around, walk back, and sit down.

SECONDARY OUTCOMES:
Fracture | 10 years
  Incidence of fracture of all parts
Radiography | After enrollment, patients will be observed annually or every 2 years for up to 10 years.
  Radiography of the sites listed below will be performed. AP views of both knees, PA vies of both wrists, and both long legs. Sites with symptoms such as pain, sites of suspected fracture, and spine (cervical, thoracic and lumber).
Nephrocalcinosis | After enrollment, patients will be observed annually or every 2 years for up to 10 years.
  The renal ultrasound will be performed and the presence and/or progression of nephrocalcinosis will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka University Hospital, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carpenter TO, Fukumoto S, Haffner D, Imel EA, Ozono K, Ishii H, Li Z, Sandilands K, Joos-Vandewalle P, Lee C, Kanematsu M, McCullough KP, Brandi ML. Advancing Patient Evidence in XLH (APEX): Baseline analysis of a global data unification program. Bone. 2025 Dec;201:117649. doi: 10.1016/j.bone.2025.117649. Epub 2025 Sep 15. PMID 40962182
- [Derived] Ito N, Kang HG, Michigami T, Namba N, Kubota T, Shintani A, Kawai R, Kabata D, Ishii H, Nishida Y, Fukumoto S, Ozono K. Prevalence of Comorbid Hyperparathyroidism and Its Association with Renal Dysfunction in Asian Patients with X-Linked Hypophosphatemic Rickets/Osteomalacia. Calcif Tissue Int. 2025 Mar 12;116(1):50. doi: 10.1007/s00223-025-01359-9. PMID 40074938
- [Derived] Kubota T, Fukumoto S, Cheong HI, Michigami T, Namba N, Ito N, Tokunaga S, Gibbs Y, Ozono K. Long-term outcomes for Asian patients with X-linked hypophosphataemia: rationale and design of the SUNFLOWER longitudinal, observational cohort study. BMJ Open. 2020 Jun 29;10(6):e036367. doi: 10.1136/bmjopen-2019-036367. PMID 32601114